CLINICAL TRIAL: NCT07101796
Title: Distribution of Mood and Personality Characteristics and Their Influence on Treatment Compliance
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Jing MA, Principal Investigator,, Peking University First Hospital
Other Study IDs: 2024432
Record Dates: First submitted 2024-12-22; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Personality; Patient Compliance; Anxiety; Depression; Continuous Positive Airway Pressure (CPAP)
Keywords: Obstructive sleep apnea; personality; patient compliance; Anxiety; depression; Continuous Positive Airway Pressure (CPAP)
MeSH Terms: conditions — Patient Compliance; Anxiety Disorders; Depression; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obstructive sleep apnea (OSA): dignosis OSA according to the sleep study (AHI>=5)
  Interventions: Device: continous positive airway pressure (CPAP)
- non-OSA: dignosis OSA according to the sleep study (AHI <5)

INTERVENTIONS:
Device: continous positive airway pressure (CPAP) — using CPAP to treat OSA
  Groups: Obstructive sleep apnea (OSA)

SUMMARY:
This study intends to investigate the personality and psychological characteristics of OSA patients using classical standard scales and obtain treatment information and adherence data through prospective follow-up to summarize the distribution characteristics of mood and personality characteristics of OSA patients and their influence on treatment adherence. A thorough understanding of OSA patient characteristics from the perspective of personality and psychological characteristics will be of great significance to the classification of OSA patients, precision treatment, and improving treatment compliance.

DETAILED DESCRIPTION:
This study will establish a prospective cohort to conduct the study in two parts.

1. Through the personality, mood, and sleep questionnaires of patients with suspected OSA and planned sleep monitoring, the differences in personality and treatment choices of the OSA population with different personality characteristics and emotional states through follow-up.
2. The above investigation and follow-up of patients in the hospital for ventilator pressure treatment were used to observe the effect of differences in personality characteristics and mood status on ventilator treatment acceptance, stress, and compliance indicators.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18~70 years old
* Suspected OSA based on symptoms such as snoring, waking at night, daytime sleepiness, or requiring OSA screening due to related conditions; or confirmed OSA patients referred for sleep monitoring or CPAP pressure titration.
* Subjects are conscious, utterly independent in behavioral and cognitive ability, and able to answer questions independently;
* The patients gave informed consent to the study and cooperated with relevant treatment and evaluation.

Exclusion Criteria:

* Age below 18 or above 70 years old
* No symptoms suggestive of OSA and no need for OSA screening; or patients without confirmed OSA
* lacking full independence in behavior and cognitive ability, unable to answer questions independently
* Patients who did not give informed consent or were unwilling to cooperate with treatment and evaluation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients with sleep disorders other than sleep disorders and respiratory disorders;
    * Patients with severe mental diseases (such as schizophrenia, bipolar disorder, paranoid mental disorders, mental retardation associated with mental disorders, mental disorders caused by epilepsy, schizoaffective disorders) and personality disorders;
      * Patients who are taking sleep-affecting medication.
        ④ Unable to cooperate with the relevant psychological scales for depression, anxiety, personality, and others.
        ⑤ Patients who have previously used or are being treated with a non-invasive ventilator.
        ⑥ Other serious somatic diseases or other conditions that may affect ventilator treatment are unsuitable for enrollment as assessed by the investigator.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09-14 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Eysenck Personality Questionnaire (EPQ) | At baseline
  This study adopted the classic short form of the Eysenck Personality Questionnaire - Revised (EPQ-R Short Scale) to assess individual personality traits across four dimensions: Psychoticism (P), Extraversion (E), Neuroticism (N), and Lie Scale (L). Each dimension consists of 12 items, with scores ranging from 0 to 12. Higher scores indicate a stronger presence of the corresponding trait. For example, a higher score on Neuroticism reflects greater emotional instability, while a higher score on Extraversion suggests a more outgoing and active personality

SECONDARY OUTCOMES:
continuous positive airway pressure (CPAP) compliance | From CPAP initiation to the 3-month follow-up
  downloading the data from the CPAP to assess average daily usage duration (in hours) and the number of days used per week. Good adherence is typically defined as using the CPAP device for at least 4 hours per night on 70% or more nights over the past 3 consecutive months.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Ma, Principal Investigator — Peking University First Hospital
Locations (1):
- Respiratory Department of Peking University First Hospital, Beijing, Beijing Municipality, China